CLINICAL TRIAL: NCT06557213
Title: Prediction of Liver Cancer Treatment Response Based on Gut Microbiota: a Cohort Study
Brief Title: a Cohort Study (Gut Microbiota and HCC)
Status: Not yet recruiting | Type: Observational
Sponsor: Xu Yong, MD (Other)
Collaborators: Nanjing Xiershou Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Xu Yong, MD, Secretary of the Party Committee, Shenzhen Third People's Hospital
Organization: Shenzhen Third People's Hospital (Other)
Other Study IDs: KY2024-176
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect patient feces、blood、urine、serum of patients at 0, 12, 24, and 48 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To analyze the predictive role of intestinal microbiota in tyrosine kinase inhibitors (TKIs) combined with immunotherapy response in patients with intermediate and advanced liver cancer.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study. Patients with intermediate and advanced hepatocellular carcinoma who meet the enrollment and exclusion criteria are judged to be unresectable after evaluation by professional physicians, and are intended to be treated with anti-angiogenic targeted drugs combined with immune checkpoint inhibitors. During the treatment according to clinical needs, stool and blood samples were taken regularly, and the treatment response of patients was judged according to RECIST V1.1 criteria, and the common adverse reactions during treatment were evaluated by the CTCAE5.0 grading system, and the relationship between intestinal microbiota and liver cancer treatment response was analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender unlimited
2. Diagnosed as HCC through pathological or clinical examination
3. BCLC Phase B or C
4. Previously without systematic treatment
5. Irremovable
6. Intended to receive targeted anti-angiogenic drugs combined with immune checkpoint inhibitors for treatment
7. ≥ 1 measurable lesion (RECIST V1.1)
8. ECOG PS 0-1
9. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Received attenuated live vaccine within 4 weeks prior to enrollment or planned during the study period
2. Active, known or suspected autoimmune diseases
3. Known history of primary immunodeficiency
4. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
5. Pregnant or lactating female patients
6. Uncontrolled concurrent diseases
7. Currently conducting clinical trials for other drugs
8. Other patients deemed unsuitable for inclusion by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational cohort study. Patients with advanced hepatocellular carcinoma who meet the enrollment and exclusion criteria, who are judged to be unresectable after evaluation by professional physicians, are planned to be treated with anti-angiogenic targeted drugs combined with immune checkpoint inhibitors, and according to the number of such patients in Shenzhen Third People's Hospital in the case year, this study intends to include 100 study subjects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective Progression-Free Survival (PFS) | Up to approximately 1 years
  To analyse the Progression-Free Survival (PFS) of patients
Objective Secondary Clinical Endpoints - Overall Growth Phase (OS) | Up to approximately 1 years
  To analyse the Secondary Clinical Endpoints - Overall Growth Phase (OS) of patients
Objective Objective Response Rate (ORR) | Up to approximately 1 years
  To exprole the Objective Response Rate (ORR) of patients
ObjectiveDuration of Response (DOR) | Up to approximately 1 years
  To analyse the Duration of Response (DOR) of patients
Diversity analysis | 0 weeks, 12 weeks, 24 weeks and 48 weeks
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Species differential analysis | 0 weeks, 12 weeks, 24 weeks and 48 weeks
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition.
Feces Metabolomics | 0 weeks, 12 weeks, 24 weeks and 48 weeks
  Changes of metabolites in feces measured by metabolomic mass spectrometry, unsupervised PCA (principal component analysis) was performed by statistics function prcomp, identified metabolites were annotated using KEGG Compound database.
Serum Metabolomics | 0 weeks, 12 weeks, 24 weeks and 48 weeks
  Changes of metabolites in serum measured by metabolomic mass spectrometry, unsupervised PCA (principal component analysis) was performed by statistics function prcomp, identified metabolites were annotated using KEGG Compound database.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Xu, Dr, Study Chair — Secretary of the Party Committee of the Shenzhen Third People's Hospital

IPD SHARING:
Plan to Share IPD: No